CLINICAL TRIAL: NCT03819998
Title: Serum Fetuin Level as a Marker in Polycystic Ovary Syndrome
Brief Title: Serum Fetuin Level in Polycystic Ovary Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aljazeera Hospital (Other)
Collaborators: Cairo University (Other); National Research Centre, Egypt (Other)
Responsible Party: Sponsor
Other Study IDs: Fetuin
Record Dates: First submitted 2019-01-25; First posted 2019-01-29 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Polycystic Ovary
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PCOS group: women who have PCOS
  Interventions: Diagnostic Test: measurement of Fetuin-A level in serum
- control group: women who donnot have PCOS
  Interventions: Diagnostic Test: measurement of Fetuin-A level in serum

INTERVENTIONS:
Diagnostic Test: measurement of Fetuin-A level in serum — Fetuin A level will be measured in blood of the PCOS women
  Other Names: Fwtuin A level

SUMMARY:
polycystic ovary syndrome is a common gynecological problem

DETAILED DESCRIPTION:
Understanding the pathophysiology and the cause is of much importance for proper management of this problem

ELIGIBILITY:
Inclusion Criteria:

* women who have PCOS in group 1 and who donnot have PCOS in group 2 with age between 20 -42 years

Exclusion Criteria:

* women above 42 years old

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women with polycystic ovary syndrome
Study Population: women who have PCOS and have symptoms of hyperandrogenism and irregular cycles
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-01-30 (Actual); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-02-05 (Estimated)

PRIMARY OUTCOMES:
The number of women who will have high level of fetuin A and has PCOS | within a week
  Evaluation of women who have PCOS in relation to fetuin A level

CONTACTS AND LOCATIONS:
Locations (1):
- Algazeerah and Kasralainy hospital, Giza, Egypt